CLINICAL TRIAL: NCT06145737
Title: HOme-Based Self-management and COgnitive Training CHanges Lives (HOBSCOTCH) - Multiple Sclerosis (MS)
Acronym: HOBSCOTCH-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elaine T. Kiriakopoulos, Assistant Professor of Neurology, Geisel School of Medicine at Dartmouth Director, HOBSCOTCH Institute for Cognitive Health & Well-Being Dartmouth Hitchcock Epilepsy Center, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02002107
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Cognitive Dysfunction; Memory Disorders
Keywords: Multiple Sclerosis; Memory Disorders; Cognition; Self-Management
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MS Participant with Cognitive Dysfunction (Other): Participants will receive the HOBSCOTCH-MS intervention consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH Session (on webcam or by phone)
  * 1 educational session (on webcam)
  * 6 HOBSCOTCH intervention sessions (webcam or phone)
  * 1 wrap-up session (webcam or phone)
  Interventions: Behavioral: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH)

INTERVENTIONS:
Behavioral: HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH) — One on one virtual self-management program for cognitive dysfunction associated with Multiple Sclerosis (MS).
  HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. HOBSCOTCH-MS is an adaptation of the HOBSCOTCH program for people with MS and incorporates education about multiple sclerosis and cognition into the education module.
  Other Names: HOBSCOTCH-MS

SUMMARY:
The goal of this pilot study is to assess the feasibility of adapting and delivering the existing home-based epilepsy self-management intervention, HOBSCOTCH, for people with multiple sclerosis (MS).

The main questions it aims to answer are:

1. Can the current HOBSCOTCH program be adapted for people with MS?
2. Will people with MS experience improved quality of life similar to that found in people with epilepsy after participating in the HOBSCOTCH program?

Participants will be asked to:

* attend nine, one-hour virtual (online and/or by telephone) HOBSCOTCH-MS sessions with a one-on-one certified HOBSCOTCH-MS coach
* complete a brief clinical questionnaire about their diagnosis of MS
* complete four questionnaires before and after the HOBSCOTCH-MS sessions about their quality of life and about memory and thinking processes
* keep a short daily diary about their MS symptoms and use of the self-management strategies taught in the HOBSCOTCH-MS program
* complete a brief Satisfaction Survey after the entire HOBSCOTCH-MS program

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 65 years
* Literate, English-speaking with grade 12 or equivalent in education
* Self-reported diagnosis of MS
* Self-reported cognitive/memory difficulties
* Telephone and internet access

Exclusion Criteria:

* Cognitive dysfunction that precludes participation in giving informed consent
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access
* Acute psychiatric illness
* History of progressive neurodegenerative disease (dementia)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as measured by comparing FAMS-Functional Assessment of Multiple Sclerosis v4.0 scores pre- and post-HOBSCOTCH-MS intervention. | Baseline (pre-HOBSCOTCH-MS) and post-HOBSCOTCH-MS, approximately 9 weeks later.
  The Functional Assessment of Multiple Sclerosis (FAMS) is a validated self-report health-related quality-of-life instrument for people with multiple sclerosis. The FAMS consists of 44 scored (5-point Likert scale) items in six quality-of-life domains: Mobility (seven items), Symptoms (seven items), Emotional wellbeing (seven items), General contentment (seven items), Thinking/fatigue (nine items), and Family/social wellbeing (seven items). An Additional concerns subscale consists of 15 other items that fall outside of the six domains but may provide valuable information to the clinician. The FAMS includes items across the International Classification of Functioning components of body functions, activities and participation, and environmental factors. Higher scores indicate better quality of life.
Change in subjective cognition as measured by comparing Neuro-QOL Item Bank v2.0 Cognitive Function scores pre- and post-HOBSCOTCH-MS intervention. | Baseline (pre-HOBSCOTCH-MS) and post-HOBSCOTCH-MS, approximately 9 weeks later.
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.

SECONDARY OUTCOMES:
Change in objective cognition as measured by comparing Symbol-Digit Modalities Test scores pre- and post-HOBSCOTCH-MS intervention. | Baseline (pre-HOBSCOTCH-MS) and post-HOBSCOTCH-MS, approximately 9 weeks later.
  The Symbol Digit Modalities Test (SDMT) is a validated tool that measures cognitive processing speed. It requires a person to substitute a number (1 - 9), either orally or written, for randomized presentations of geometric figures over 90 seconds. Scores range between 0 and 100 with a lower score representing poorer performance.
Change in objective cognition as measured by comparing California Verbal Learning Test-III scores pre- and post-HOBSCOTCH-MS intervention. | Baseline (pre-HOBSCOTCH-MS) and post-HOBSCOTCH-MS, approximately 9 weeks later.
  The California Verbal Learning Test-III is a validated verbal learning and memory assessment. It consists of a 16-word, list-recall task with up to five learning/recall trials. Higher scores of recall over time are associated with better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Kiriakopoulos, MD, MPH, MSc, Principal Investigator — Dartmouth-Hitchcock Medical Center; Heather A Wishart, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No